CLINICAL TRIAL: NCT04603014
Title: Initial Feasibility Pilot Study of Interdialytic Peritoneal Ultrafiltration to Manage Volume Status in Hemodialysis Patients
Brief Title: Interdialytic Peritoneal UltraFiltration in HemoDialysis Patients
Acronym: IPUF-HD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Sequana Medical N.V. (Industry)
Responsible Party: Principal Investigator, Chris McIntyre, Professor of Medicine, Medical Biophysics and Pediatrics, School of Medicine and Dentistry, Western University; Director of The Kidney Clinical Research Unit, London Health Sciences Centre, London, ON, Canada, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115423
Record Dates: First submitted 2020-10-13; First posted 2020-10-26 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: End Stage Renal Disease on Dialysis; Hemodialysis; Peritoneal Dialysis; Nonosmotic Sodium Storage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interdialytic peritoneal ultrafiltration (Experimental): Will receive incremental interdialytic peritoneal ultrafiltration with a 10% dextrose solution, twice a week for three consecutive weeks
  Interventions: Combination Product: Interdialytic peritoneal ultrafiltration with 10% dextrose solution

INTERVENTIONS:
Combination Product: Interdialytic peritoneal ultrafiltration with 10% dextrose solution — Interdialytic peritoneal ultrafiltration with incremental doses of a 10% dextrose solution, after hemodialysis twice weekly for three consecutive weeks

SUMMARY:
Sodium accumulates in the tissues of patients with kidney disease and impairs survival. Three-times weekly, standard hemodialysis alone cannot remove excess sodium efficiently. A sample of 10 chronic hemodialysis patients will undergo a 5-week, pilot, interventional study to test the efficacy of additional sodium removal in-between hemodialysis sessions, twice per week, for three weeks. Tissue sodium removal will be achieved with peritoneal dialysis after the surgical insertion of a peritoneal dialysis catheter. Tissue sodium removal will be assessed at the beginning and at the end of the study with sodium magnetic resonance imaging of a peripheral limb (leg). Patients will also undergo monitoring for symptoms and blood pressure throughout the study to assess the safety of this procedure.

DETAILED DESCRIPTION:
Hypothesis: Interdialytic peritoneal ultrafiltration (iPUF) via Tenckhoff peritoneal dialysis catheter using 10% Dextrose infusate is feasible and provides effective volume management and sodium removal in prevalent HD patients.

Overview: This is a prospective, interventional pilot study from the London Health Sciences Centre (LHSC) prevalent HD population. Study patients will undergo the surgical implantation of a Tenckhoff peritoneal dialysis catheter before study start. After the successful insertion of the Tenckhoff catheter, study patients will enter a run-in phase, where their residual renal function, volume, hemodynamic and cardiac status during HD will be assessed. During the following weeks (intervention weeks 1, 2, 3), study patients will receive in-center iPUF intervention, consisting of peritoneal infusate instillation of a 10% dextrose solution via a Tenckhoff catheter, immediately after the first two HD sessions of the week (Monday, Wednesday); the infusate will be dwelling in the study patient's peritoneal cavity for 2 hours, at the end of which the solution will be drained and the patient sent home. Study patients will be monitored during infusate administration and for the first four hours thereafter. The study intervention will be discontinued at the beginning of week 5 (Wash-out); during week 5 and the first HD session of week 6, study patients will be monitored to observe potential residual effects of the iPUF intervention.

ELIGIBILITY:
Inclusion Criteria

* At least one of the following:

  * Average per-session interdialytic weight gain ≥ 4.0 % of their dry weight in the last month;
  * Inability to consistently achieve dry weight with the current treatment schedule;
  * Need for additional HD treatments to achieve prescribed dry weight.
* Weekly HD sessions - up to three times/week
* Age ≥18 years
* Willing and able to give informed consent

Exclusion Criteria

* Contraindications to peritoneal dialysis
* Contraindications to MRI
* Uncontrolled diabetes mellitus
* Active infections
* Non-compliance to hemodialysis prescription
* Pre-study serum sodium < 130 mmol/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Skin sodium concentration | End of week 4
  Skin sodium concentration at the end of week 4 as measured by sodium-23 magnetic resonance imaging of the leg.
Adverse events | iPUF interventions on Week 2, 3 and 4
  Completion of the iPUF treatment without adverse events

SECONDARY OUTCOMES:
Interdialytic weight gain | week 1 vs 4, week 1 vs 5-6
  Difference in interdialytic weight gain at run-in week vs end of intervention, vs wash-out
Total weekly sodium removal with interdialytic peritoneal ultrafiltration | week 2, 3, 4
  Total weekly sodium removal with peritoneal dialysis in intervention weeks
Total volume of fluid removed with interdialytic peritoneal ultrafiltration | week 2, 3, 4
  Total volume of fluid removed with peritoneal dialysis in intervention weeks
Home blood pressure | week 1 vs week 4, week 1 vs 5-6
  Changes in home blood pressure at baseline vs end of intervention and vs washout
Mean intradialytic hemodynamics | week 1 vs 4, week 1 vs 6
  Changes in mean intradialytic hemodynamic monitor parameters, as measured with Finometer and CVInsight
Regional wall motion abnormalities | week 1 vs 4, week 1 vs 6
  Changes in Regional Wall Motion Abnormalities (echocardiography) at peak-stress hemodialysis
Symptoms | week 1 vs 4, week 1 vs 6
  Changes in symptoms as measured with the London Evaluation of Illness questionnaire
Infusion pain | Through study completion, average of all study treatments
  Infusion pain as measured with 0-10 visual analog scale
Changes in serum sodium | Through study completion, average of all study treatments
  Post-iPUF change in serum sodium

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W. McIntyre, MD, PhD, Principal Investigator — Lawson Research Institute
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flythe JE, Curhan GC, Brunelli SM. Disentangling the ultrafiltration rate-mortality association: the respective roles of session length and weight gain. Clin J Am Soc Nephrol. 2013 Jul;8(7):1151-61. doi: 10.2215/CJN.09460912. Epub 2013 Mar 14. PMID 23493384
- [Background] Assimon MM, Wang L, Flythe JE. Failed Target Weight Achievement Associates with Short-Term Hospital Encounters among Individuals Receiving Maintenance Hemodialysis. J Am Soc Nephrol. 2018 Aug;29(8):2178-2188. doi: 10.1681/ASN.2018010004. Epub 2018 May 23. PMID 29793962
- [Background] Ramdeen G, Tzamaloukas AH, Malhotra D, Leger A, Murata GH. Estimates of interdialytic sodium and water intake based on the balance principle: differences between nondiabetic and diabetic subjects on hemodialysis. ASAIO J. 1998 Nov-Dec;44(6):812-7. doi: 10.1097/00002480-199811000-00009. PMID 9831090
- [Background] Titze J, Lang R, Ilies C, Schwind KH, Kirsch KA, Dietsch P, Luft FC, Hilgers KF. Osmotically inactive skin Na+ storage in rats. Am J Physiol Renal Physiol. 2003 Dec;285(6):F1108-17. doi: 10.1152/ajprenal.00200.2003. Epub 2003 Jul 29. PMID 12888617
- [Background] Kopp C, Linz P, Wachsmuth L, Dahlmann A, Horbach T, Schofl C, Renz W, Santoro D, Niendorf T, Muller DN, Neininger M, Cavallaro A, Eckardt KU, Schmieder RE, Luft FC, Uder M, Titze J. (23)Na magnetic resonance imaging of tissue sodium. Hypertension. 2012 Jan;59(1):167-72. doi: 10.1161/HYPERTENSIONAHA.111.183517. Epub 2011 Dec 5. PMID 22146510
- [Background] Machnik A, Neuhofer W, Jantsch J, Dahlmann A, Tammela T, Machura K, Park JK, Beck FX, Muller DN, Derer W, Goss J, Ziomber A, Dietsch P, Wagner H, van Rooijen N, Kurtz A, Hilgers KF, Alitalo K, Eckardt KU, Luft FC, Kerjaschki D, Titze J. Macrophages regulate salt-dependent volume and blood pressure by a vascular endothelial growth factor-C-dependent buffering mechanism. Nat Med. 2009 May;15(5):545-52. doi: 10.1038/nm.1960. Epub 2009 May 3. PMID 19412173
- [Background] Wenstedt EFE, Olde Engberink RHG, Vogt L. Sodium Handling by the Blood Vessel Wall: Critical for Hypertension Development. Hypertension. 2018 Jun;71(6):990-996. doi: 10.1161/HYPERTENSIONAHA.118.10211. Epub 2018 Apr 16. No abstract available. PMID 29661837
- [Background] Qirjazi E, Salerno FR, Akbari A, Hur L, Penny J, Scholl T, McIntyre CW. Tissue sodium concentrations in chronic kidney disease and dialysis patients by lower leg sodium-23 magnetic resonance imaging. Nephrol Dial Transplant. 2020 Apr 6:gfaa036. doi: 10.1093/ndt/gfaa036. Online ahead of print. PMID 32252091
- [Background] Canaud B, Kooman J, Selby NM, Taal M, Francis S, Kopperschmidt P, Maierhofer A, Kotanko P, Titze J. Sodium and water handling during hemodialysis: new pathophysiologic insights and management approaches for improving outcomes in end-stage kidney disease. Kidney Int. 2019 Feb;95(2):296-309. doi: 10.1016/j.kint.2018.09.024. PMID 30665570
- [Background] Dahlmann A, Dorfelt K, Eicher F, Linz P, Kopp C, Mossinger I, Horn S, Buschges-Seraphin B, Wabel P, Hammon M, Cavallaro A, Eckardt KU, Kotanko P, Levin NW, Johannes B, Uder M, Luft FC, Muller DN, Titze JM. Magnetic resonance-determined sodium removal from tissue stores in hemodialysis patients. Kidney Int. 2015 Feb;87(2):434-41. doi: 10.1038/ki.2014.269. Epub 2014 Aug 6. PMID 25100048
- [Background] Santos SF, Peixoto AJ. Sodium balance in maintenance hemodialysis. Semin Dial. 2010 Nov-Dec;23(6):549-55. doi: 10.1111/j.1525-139X.2010.00794.x. PMID 21175831
- [Background] Obi Y, Rhee CM, Mathew AT, Shah G, Streja E, Brunelli SM, Kovesdy CP, Mehrotra R, Kalantar-Zadeh K. Residual Kidney Function Decline and Mortality in Incident Hemodialysis Patients. J Am Soc Nephrol. 2016 Dec;27(12):3758-3768. doi: 10.1681/ASN.2015101142. Epub 2016 May 11. PMID 27169576
- [Background] Kawanishi H, Hashimoto Y, Nakamoto H, Nakayama M, Tranaeus A. Combination therapy with peritoneal dialysis and hemodialysis. Perit Dial Int. 2006 Mar-Apr;26(2):150-4. No abstract available. PMID 16623416
- [Background] McIntyre CW. Bimodal dialysis: an integrated approach to renal replacement therapy. Perit Dial Int. 2004 Nov-Dec;24(6):547-53. PMID 15559484
- [Background] Sriperumbuduri S, Biyani M, Brown PA, McCormick BB. Retrospective study of patients on hybrid dialysis: Single-center data from North America. Perit Dial Int. 2020 Mar;40(2):224-226. doi: 10.1177/0896860819887284. Epub 2020 Jan 17. PMID 32063198
- [Background] Banshodani M, Kawanishi H, Moriishi M, Shintaku S, Tsuchiya S. Association between Dialysis Modality and Cardiovascular Diseases: A Comparison between Peritoneal Dialysis and Hemodialysis. Blood Purif. 2020;49(3):302-309. doi: 10.1159/000504040. Epub 2019 Dec 18. PMID 31851981
- [Background] Kanda R, Io H, Nakata J, Makita Y, Sasaki Y, Matsumoto M, Wakabayashi K, Tomino Y, Suzuki Y. Evaluation of Long-Term Combination Therapy With Peritoneal Dialysis and Hemodialysis. Ther Apher Dial. 2017 Apr;21(2):180-184. doi: 10.1111/1744-9987.12517. Epub 2017 Feb 10. PMID 28185405
- [Background] Rao VS, Turner JM, Griffin M, Mahoney D, Asher J, Jeon S, Yoo PS, Boutagy N, Feher A, Sinusas A, Wilson FP, Finkelstein F, Testani JM. First-in-Human Experience With Peritoneal Direct Sodium Removal Using a Zero-Sodium Solution: A New Candidate Therapy for Volume Overload. Circulation. 2020 Mar 31;141(13):1043-1053. doi: 10.1161/CIRCULATIONAHA.119.043062. Epub 2020 Jan 8. PMID 31910658
- [Background] Quiroga IM, Baboo R, Lord RH, Darby CR. Tenckhoff catheters post-renal transplantation: the 'pull' technique? Nephrol Dial Transplant. 2001 Oct;16(10):2079-81. doi: 10.1093/ndt/16.10.2079. PMID 11572901
- [Background] Grieff M, Mamo E, Scroggins G, Kurchin A. The 'Pull' Technique for Removal of Peritoneal Dialysis Catheters: A Call for Re-Evaluation of Practice Standards. Perit Dial Int. 2017 Mar-Apr;37(2):225-229. doi: 10.3747/pdi.2016.00152. PMID 28360368
- [Background] Quiroga I, Reddy SP, Bhattacharjya S, Darby CR. Tenckhoff catheters: the pull technique. Nephrol Dial Transplant. 2003 Aug;18(8):1682. doi: 10.1093/ndt/gfg173. No abstract available. PMID 12897121
- [Derived] McIntyre CW. Update on Hemodialysis-Induced Multiorgan Ischemia: Brains and Beyond. J Am Soc Nephrol. 2024 May 1;35(5):653-664. doi: 10.1681/ASN.0000000000000299. Epub 2024 Jan 26. PMID 38273436